CLINICAL TRIAL: NCT01168401
Title: Phase 1, Randomized Controlled Dose Escalation, Safety and Immunogenicity Study of Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-Like Particle (VLP) Vaccine Adjuvanted With Monophosphoryl Lipid A (MPL) and Aluminum Hydroxide [Al(OH)3] in Adults
Brief Title: Bivalent Norovirus Vaccine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LV03-104; U1111-1187-1052 (Registry Identifier: WHO)
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-04

CONDITIONS: Gastroenteritis
Keywords: Vaccine, norovirus, acute gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NoV GI.1/GII.4 Bivalent VLP Vaccine (Experimental): Norovirus Bivalent GI.1 and GII.4 VLP Vaccine, adjuvanted with 50 microgram (mcg) MPL and 500 mcg Al(OH)3, IM, on Days 0 and 28.
  Interventions: Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine
- Saline (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: NoV GI.1/GII.4 Bivalent VLP Vaccine — 2 Doses 28 days apart Cohort A: 18-49 Years
  Cohort A1: IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (5/5 mcg)
  Cohort A2: IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (15/15 mcg)
  Cohort A3: IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (50/50 mcg)
  Cohort A4: IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (150/150 mcg)
  Cohort B: 50-64 Years IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (50/50 mcg)
  Cohort C: 65-85 Years IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (50/50 mcg)
  Cohort D: 18-49 Years IM Norovirus Bivalent GI.1/GII.4 VLP Vaccine (50/50 mcg)
  Arms: NoV GI.1/GII.4 Bivalent VLP Vaccine
Biological: Saline — Two doses 28 days apart
  Arms: Saline

SUMMARY:
Randomized, multi-site, dose-escalation study of the safety and immunogenicity of four dosage levels of Intramuscular (IM) Norovirus Bivalent VLP Vaccine adjuvanted with MPL and Al(OH)3 compared to controls. Participants will receive two doses, by IM injection, 28 days apart.

The hypotheses for this study are:

* The incidence of adverse events after vaccination with IM Norovirus Bivalent VLP Vaccine will be similar to the incidence of adverse events after other IM vaccines including CERVARIX® which contains MPL and Al(OH)3.
* Two doses of IM Norovirus Bivalent VLP Vaccine will be more immunogenic than one dose.
* The post-vaccination serum antibody responses, the number of antibody secreting cells (ASC), including homing markers, and memory B-cell responses directed against norovirus antigens will be increased after IM Norovirus Bivalent VLP Vaccine compared to controls.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria listed below:

1. Signed written informed consent.
2. Age:

   * Cohort A: 18-49 years, inclusive
   * Cohort B: 50-64 years, inclusive
   * Cohort C: 65-85 years, inclusive
   * Cohort D: 18-49 years, inclusive
3. Health Status:

   * Cohort A and D: In good health as determined by a screening evaluation that includes vital signs, medical history, and physical exam within 45 days before administration of IM Norovirus Bivalent VLP Vaccine or control.
   * Cohorts B and C: In good health as determined by a screening evaluation that includes vital signs, medical history, and physical exam within 45 days before administration of IM Norovirus Bivalent VLP Vaccine or control. Any existing medical diagnoses or conditions must be stable based on medical history and targeted physical examination. A stable medical condition is defined as: (A) Clinically acceptable health outcomes for the specific condition over the prior 6 months and (B) No change in prescription medication(s), dose, or frequency over the prior 3 months. Acceptable changes in medications are: a change of health care provider or insurance company or that is made for financial reasons as long as the medications are in the same class and/or a change due to improvement in a disease outcome.
4. Expressed interest and availability to fulfill the study requirements.
5. Female participants must be of non-childbearing potential (surgically sterile or post-menopausal for greater than or equal to [>=] 12 months), or if of childbearing potential (as determined by the investigator) must be practicing abstinence or using an effective licensed method of birth control (example oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream, or foam; intrauterine contraceptive device, or Depo-Provera; skin patch; vaginal ring or cervical cap) for 30 days prior to vaccination and must agree to continue such precautions for at least 60 days after the last vaccination. A woman is eligible if she is monogamous with a male who has had a vasectomy. Male participants must agree not to father a child for at least 60 days after the last vaccination and to practice abstinence or use an effective method of birth control as noted above.
6. Agrees not to participate in another clinical trial with an investigational product for the entire duration of the study one year after the last study dose that is 393 days.
7. Agrees to storage of unused clinical specimens for an indefinite period of time for future norovirus research or research on other gastrointestinal pathogens.

Exclusion Criteria:

Participants who meet any of the exclusion criteria at baseline will be excluded from study participation. The exclusion criteria are:

1. History of any of the following medical illnesses:

   * Diabetes
   * Cancer (malignancy other than resolved/excised skin lesion)
   * Heart disease (hospitalization for a heart attack, arrhythmia, or syncope)
   * Unconsciousness (other than a single brief "concussion")
   * Seizures (other than febrile seizures as a child less than [<] 5 years old)
   * Recurrent infections (more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
   * Any condition associated with immunodeficiency or participants taking immunosuppressant medication
   * Neuroinflamatory or auto-immune disease
2. Any current illness requiring daily medication other than the following:

   * Cohort A and D: Vitamins, birth control, anti-hypertensive medication, antihistamines or anti-depressant medication. The Principal Investigator (PI) should consult with the Central Safety Monitor and/or the sponsor for any clarification of medications allowable.
   * Cohorts B and C: Vitamins, birth control, anti-hypertensive medication, antihistamines or anti-depressant medication or any current illness requiring daily medication other than as noted above in inclusion criteria 3. The PI should consult with the Central Safety Monitor and/or the sponsor for any clarification of medications allowable.
3. Allergies or hypersensitivity to any component of the vaccine including MPL and Al(OH)3 adjuvants.
4. Any clinically significant abnormality detected on physical examination, including:

   * Murmur (other than a functional murmur)
   * Focal neurological abnormality
   * Hepatosplenomegaly
   * Lymphadenopathy
   * Jaundice
5. Hypertension (Blood Pressure [BP] greater than [>] 140/90 millimeter of mercury [mm Hg] on two separate days)
6. Any lab abnormality (per the site local laboratory), as listed below:

   * Absolute Neutrophil Count (ANC) outside the normal range (may be repeated if outside this limit)
   * Total white blood cells (WBC) outside the normal range (may be repeated if outside this limit)
   * Hemoglobin outside the normal range (may be repeated if outside this limit)
   * Platelet count outside the normal range (may be repeated if outside this limit)
   * Blood urea nitrogen (BUN) > upper limit of normal (ULN) (may be repeated if outside this limit)
   * Creatinine > ULN (may be repeated if outside this limit)
   * Glucose (fasting or random) outside the normal range (may be repeated if outside this limit)
   * Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) > ULN (may be repeated if outside this limit)
7. Positive serology for hepatitis C or Human Immunodeficiency Virus (HIV) antibody or hepatitis B surface antigen.
8. For women of child bearing potential, positive serum pregnancy test within 14 days and urine pregnancy test within 24 hours of administering either dose of IM Norovirus Bivalent VLP Vaccine or control.
9. Nursing mother.
10. Temperature >100.4 degree Fahrenheit (F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 3 days of administration of IM Norovirus Bivalent VLP Vaccine or control.
11. Previous participation in a Norovirus vaccine or challenge study.
12. Study site personnel or their family members.
13. Significant history of psychiatric hospitalization, alcohol abuse, or illicit drug use in the prior 5 years.
14. Completion of an investigational vaccine or drug study within 28 days before administration of IM Norovirus Bivalent VLP Vaccine or control.
15. Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
16. Other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a participant participating in the trial, would render the participant unable to comply with the protocol or would interfere with the evaluation of the vaccine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-09-03 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Navy Medical Research Center, Silver Springs, Maryland
  - Saint Louis University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Derived] Ramani S, Neill FH, Ferreira J, Treanor JJ, Frey SE, Topham DJ, Goodwin RR, Borkowski A, Baehner F, Mendelman PM, Estes MK, Atmar RL. B-Cell Responses to Intramuscular Administration of a Bivalent Virus-Like Particle Human Norovirus Vaccine. Clin Vaccine Immunol. 2017 May 5;24(5):e00571-16. doi: 10.1128/CVI.00571-16. Print 2017 May. PMID 28249841
- [Derived] Lindesmith LC, Ferris MT, Mullan CW, Ferreira J, Debbink K, Swanstrom J, Richardson C, Goodwin RR, Baehner F, Mendelman PM, Bargatze RF, Baric RS. Broad blockade antibody responses in human volunteers after immunization with a multivalent norovirus VLP candidate vaccine: immunological analyses from a phase I clinical trial. PLoS Med. 2015 Mar 24;12(3):e1001807. doi: 10.1371/journal.pmed.1001807. eCollection 2015 Mar. PMID 25803642
- [Derived] Treanor JJ, Atmar RL, Frey SE, Gormley R, Chen WH, Ferreira J, Goodwin R, Borkowski A, Clemens R, Mendelman PM. A novel intramuscular bivalent norovirus virus-like particle vaccine candidate--reactogenicity, safety, and immunogenicity in a phase 1 trial in healthy adults. J Infect Dis. 2014 Dec 1;210(11):1763-71. doi: 10.1093/infdis/jiu337. Epub 2014 Jun 20. PMID 24951828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 03 September 2010 to 09 January 2013.
Pre-assignment Details: Healthy volunteers were enrolled in 1 of the following treatment groups: Bivalent Norovirus GI.1/GII.4 Vaccine (Cohort A: 5/5 microgram [mcg], 15/15 mcg, 50/50 mcg, 150/150 mcg; Cohort B: 50/50 mcg; Cohort C: 50/50 mcg and Cohort D: 50/50 mcg) adjuvanted with 50 mcg monophosphoryl lipid A (MPL) and 500 mcg aluminum hydroxide [Al(OH)3]) or Placebo.
Groups:
- Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg: Norovirus bivalent Virus-Like Particle (VLP) Vaccine (5 mcg of GI.1 norovirus VLP and 5 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A2:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg: Norovirus bivalent VLP Vaccine (15 mcg of GI.1 norovirus VLP and 15 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg; Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg: Norovirus bivalent VLP Vaccine (50 mcg of GI.1 norovirus VLP and 50 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg: Norovirus bivalent VLP Vaccine (150 mcg of GI.1 norovirus VLP and 150 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A1-A4: Placebo: Norovirus Bivalent VLP Placebo-matching injection (0.9 percent [%] sodium chloride [NaCl] and preservative-free), intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg: Norovirus bivalent VLP Vaccine (50 mcg of GI.1 norovirus VLP and 50 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 50-64 years.
- Cohort B: Placebo: Norovirus Bivalent VLP Placebo-matching injection (0.9% NaCl and preservative-free), intramuscularly, on Days 0 and 28 in participants aged 50-64 years.
- Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg: Norovirus bivalent VLP Vaccine (50 mcg of GI.1 norovirus VLP and 50 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 65-85 years.
- Cohort C: Placebo: Norovirus Bivalent VLP Placebo-matching injection (0.9% NaCl and preservative-free), intramuscularly, on Days 0 and 28 in participants aged 65-85 years.
- Cohort D: Placebo: Norovirus Bivalent VLP Placebo-matching injection (0.9% NaCl and preservative-free), intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
Period: Overall Study
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Started | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
Completed | 9 | 9 | 8 | 7 | 9 | 9 | 10 | 10 | 9 | 8 | 8
Not Completed | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) population included all participants who received at least 1 dose of study product.
Groups:
- Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg: Norovirus bivalent VLP Vaccine (5 mcg of GI.1 norovirus VLP and 5 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg: Norovirus bivalent VLP Vaccine (15 mcg of GI.1 norovirus VLP and 15 mcg of GII.4 norovirus VLP) adjuvanted with 50 mcg MPL and 500 mcg Al(OH)3, injection, intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Cohort A1-A4: Placebo; Cohort D: Placebo: Norovirus Bivalent VLP Placebo-matching injection (0.9% NaCl and preservative-free), intramuscularly, on Days 0 and 28 in participants aged 18-49 years.
- Total: Total of all reporting groups
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8 | 102
Age, Customized [Number; unit: participants]
  Greater than or equal to (>=) 18 and <64 years | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 0 | 0 | 8 | 8 | 83
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9 | 0 | 0 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 7 | 8 | 5 | 5 | 8 | 5 | 3 | 7 | 68
  Male | 3 | 4 | 3 | 2 | 1 | 4 | 5 | 2 | 4 | 5 | 1 | 34
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8 | 102
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Black or African American | 2 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 5 | 5 | 19
  White | 8 | 7 | 6 | 6 | 7 | 9 | 9 | 10 | 9 | 3 | 2 | 76
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Ethnicity [Count of Participants; unit: Participants]
  Non-Hispanic | 8 | 10 | 10 | 9 | 9 | 9 | 9 | 10 | 9 | 6 | 8 | 97
  Hispanic | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5
Saliva Secretor Status [Count of Participants; unit: Participants]
  Saliva Secretor Status Positive | 7 | 8 | 6 | 9 | 8 | 6 | 8 | 8 | 7 | 7 | 5 | 79
  Saliva Secretor Status Negative | 3 | 2 | 4 | 0 | 1 | 3 | 2 | 2 | 2 | 1 | 3 | 23
Blood Type [Count of Participants; unit: Participants]
  Blood Type A | 3 | 3 | 5 | 3 | 2 | 2 | 6 | 3 | 2 | 1 | 2 | 32
  Blood Type B | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 2 | 2 | 11
  Blood Type O | 6 | 4 | 5 | 5 | 5 | 5 | 3 | 7 | 5 | 5 | 3 | 53
  Blood Type AB | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) Post Dose 1
Description: The solicited local adverse events were reported using a memory aid. Pain was scaled as Mild (did not interfere with activity); Moderate (repeated use of non-narcotic pain reliever greater than (>) 24 hours [24h] or interfered with activity); and Severe (any use of narcotic pain reliever or prevented daily activity). Tenderness was scaled as Mild (mild discomfort to touch); Moderate (discomfort with movement); and Severe (significant discomfort at rest). Swelling and redness were scaled as Mild (2.5-5 centimeter [cm] and did not interfere with activity); Moderate (5.1-10 cm or interfered with activity); and Severe (>10 cm or prevented daily activity).
Time Frame: Day 0 up to Day 7
Population: mITT population included all participants who received at least 1 dose of study product. Only those categories have been reported below where at least 1 participant experienced the event.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
participants
  Pain: Mild | 4 | 5 | 6 | 5 | 1 | 5 | 0 | 4 | 0 | 4 | 0
  Pain: Moderate | 4 | 2 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Tenderness: Mild | 4 | 5 | 6 | 5 | 1 | 4 | 1 | 6 | 0 | 3 | 2
  Tenderness: Moderate | 3 | 4 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Swelling: Mild | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 3 | 3

2. Primary Outcome: Number of Participants With Solicited Local AEs Post Dose 2
Description: The solicited local adverse events were reported using a memory aid. Pain was scaled as Mild (did not interfered with activity); Moderate (repeated use of non-narcotic pain reliever >24h or interfered with activity); and Severe (any use of narcotic pain reliever or prevented daily activity). Tenderness was scaled as Mild (mild discomfort to touch); Moderate (discomfort with movement); and Severe (significant discomfort at rest). Swelling and redness were scaled as Mild (2.5-5 cm and did not interfere with activity); Moderate (5.1-10 cm or interfered with activity); and Severe (>10 cm or prevented daily activity).
Time Frame: Day 28 up to Day 35
Population: mITT population where Day 28 to 35 assessment were available for this measure. mITT population included all participants who received at least 1 dose of study product. Only those categories have been reported below where at least 1 participant experienced the event.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
participants
  Pain: Mild | 5 | 4 | 4 | 2 | 0 | 3 | 0 | 5 | 0 | 3 | 1
  Pain: Moderate | 3 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
  Tenderness: Mild | 7 | 6 | 6 | 3 | 1 | 6 | 1 | 4 | 0 | 5 | 2
  Tenderness: Moderate | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Swelling: Mild | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 5
  Swelling: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Mild | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic AEs Post Dose 1
Description: Elevated oral temperature:Mild(38-38.4 Celsius[C]);Moderate(38.5-38.9 C);Severe(39-40 C).Headache:Mild(no interference with activity);Moderate(repeated use of non-narcotic pain reliever>24h/some interference with activity);Severe(significant;any use of narcotic pain reliever/prevented daily activity).Fatigue,Malaise:Mild(no interference with activity);Moderate(some interference with activity);Severe(significant;prevented daily activity).Diarrhea:Mild(2-3loose stools/<400gram[g]/24h);Moderate(4-5stools/400-800g/24h);Severe(>=6watery stools/>800g/24h/required intravenous[IV]hydration).Nausea/Vomiting:Mild(no interference with activity/1-2 episodes/24h);Moderate(some interference with activity/>2 episodes/24h);Severe(prevented daily activity,required IV hydration).Muscle ache,chills,joint ache,abdominal cramp/pain:Mild(no interference with activity);Moderate(some interference with activity,not required medical intervention);Severe(prevented daily activity,required medical intervention).
Time Frame: Day 0 up to Day 7
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
participants
  Headache: Mild | 1 | 3 | 3 | 2 | 2 | 5 | 0 | 2 | 2 | 0 | 2
  Headache: Moderate | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Fatigue/ Malaise: Mild | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Fatigue/ Malaise: Moderate | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Aches : Mild | 4 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Aches : Moderate | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Joint Aches: Mild | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Aches: Moderate | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Mild | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
  Nausea: Moderate | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal Cramps/Discomfort: Mild | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Abdominal Cramps/Discomfort: Moderate | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Chills: Mild | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Moderate | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea: Mild | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
  Diarrhea: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Diarrhea: Severe | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Solicited Systemic AEs Post Dose 2
Description: Elevated oral temperature:Mild(38-38.4 C);Moderate(38.5-38.9 C);Severe(39-40 C).Headache:Mild(no interference with activity);Moderate(repeated use of non-narcotic pain reliever>24h/some interference with activity);Severe(significant;any use of narcotic pain reliever/prevented daily activity).Fatigue,Malaise:Mild(no interference with activity);Moderate(some interference with activity);Severe(significant;prevented daily activity).Diarrhea:Mild(2-3loose stools/<400g/24h);Moderate(4-5stools/400-800g/24h);Severe(>=6watery stools/>800g/24h/required IV hydration).Nausea/Vomiting:Mild(no interference with activity/1-2 episodes/24h);Moderate(some interference with activity/>2 episodes/24h);Severe(prevented daily activity,required IV hydration).Muscle ache,chills,joint ache,abdominal cramp/pain:Mild(no interference with activity);Moderate(some interference with activity,not required medical intervention);Severe(prevented daily activity,required medical intervention).
Time Frame: Day 28 up to Day 35
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
participants
  Headache: Mild | 1 | 1 | 3 | 2 | 1 | 3 | 0 | 1 | 1 | 1 | 1
  Headache: Moderate | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Fatigue/ Malaise: Mild | 1 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Fatigue/ Malaise: Moderate | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Muscle Aches: Mild | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Aches: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Joint Aches: Mild | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Joint Aches: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Nausea: Mild | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Nausea: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Abdominal Cramps/Discomfort: Mild | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Chills: Mild | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Diarrhea: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Unsolicited AEs Post Dose 1
Time Frame: Baseline up to Day 28 (Pre-dose 2)
Population: mITT population included all participants who received at least 1 dose of study product.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
participants | 7 | 4 | 4 | 1 | 2 | 4 | 0 | 3 | 3 | 3 | 4

6. Primary Outcome: Number of Participants With Unsolicited AEs Post Dose 2
Time Frame: Day 28 up to Day 56 (Post dose 2)
Population: mITT population where Day 28 to 56 assessment were available for this measure. mITT population included all participants who received at least 1 dose of study product.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
participants | 2 | 1 | 2 | 2 | 2 | 3 | 3 | 2 | 2 | 3 | 1

7. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Markedly Abnormal Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values (serum chemistry or hematology) collected throughout study.
Time Frame: Baseline up to Day 35
Population: mITT population included all participants who received at least 1 dose of study product.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
participants | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), Onset of Significant New Medical Conditions, Including Adverse Events of Special Interest (AESI)
Time Frame: Baseline up to 365 Days after post dose 2 (Day 393)
Population: mITT population included all participants who received at least 1 dose of study product.
Measure: Number; unit: participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9 | 9 | 10 | 10 | 9 | 8 | 8
participants
  SAE | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
  New Medical Conditions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Geometric Mean Titer (GMT) of Serum Anti-norovirus GI.1 and GII.4 VLP Ig (Immunoglobulin) A
Description: Run I was defined as the initial analysis performed once Day 56 post dose data was available. Run II was defined as final analysis performed after all later time points were achieved.
Time Frame: First (I) run: predose 1 and 7, 21, 28 days postdose (PD)1, and 7 and 28 days PD2; second (II) run: predose 1 and 28, 152 and 365 days PD2 (up to Day 393)
Population: Per Protocol (PP) population included all participants who received both doses of study product and with no protocol deviations likely to affect the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 9 | 9 | 8 | 7
titer
  GI.1: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run: Pre-Dose 1 | 9 [3 to 26] | 5 [3 to 7] | 5 [3 to 10] | 6 [3 to 13] | 10 [3 to 32] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 5 [3 to 8] | 5 [3 to 9] | 4 [3 to 5] | 3 [3 to 3] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 204 [126 to 332] | 357 [141 to 906] | 458 [97 to 2154] | 675 [136 to 3334] | 7 [2 to 20] | 357 [110 to 1158] | 5 [3 to 8] | 208 [48 to 903] | 4 [3 to 5] | 40 [13 to 120] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 164 [87 to 311] | 164 [71 to 379] | 269 [90 to 799] | 307 [84 to 1115] | 9 [3 to 26] | 252 [151 to 421] | 5 [3 to 9] | 114 [31 to 423] | 4 [3 to 5] | 31 [10 to 96] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:28 Days PD1 | 143 [70 to 293] | 106 [42 to 267] | 183 [61 to 544] | 149 [43 to 517] | 9 [3 to 23] | 178 [95 to 335] | 5 [3 to 8] | 104 [29 to 375] | 4 [3 to 5] | 21 [7 to 60] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 134 [62 to 291] | 112 [46 to 275] | 130 [57 to 294] | 131 [45 to 376] | 11 [3 to 34] | 140 [73 to 270] | 5 [3 to 8] | 105 [33 to 329] | 4 [3 to 5] | 19 [7 to 55] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 115 [55 to 243] | 80 [28 to 224] | 70 [24 to 202] | 78 [20 to 310] | 10 [3 to 29] | 97 [48 to 198] | 5 [3 to 8] | 76 [23 to 251] | 4 [3 to 5] | 17 [7 to 42] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:Pre-Dose 1 | 5 [2 to 9] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 3 [3 to 4] | 6 [2 to 18] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 6 [3 to 12] | 6 [3 to 13] | 5 [3 to 9] | 4 [2 to 6] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 32 [13 to 81] | 15 [7 to 33] | 11 [6 to 21] | 16 [6 to 43] | 6 [2 to 18] | 120 [62 to 231] | 6 [3 to 11] | 154 [68 to 348] | 5 [3 to 8] | 35 [13 to 99] | 3 [3 to 5]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 17 [6 to 47] | 13 [6 to 26] | 10 [6 to 19] | 16 [6 to 43] | 6 [2 to 18] | 57 [36 to 92] | 6 [3 to 12] | 78 [42 to 143] | 6 [4 to 10] | 24 [10 to 58] | 3 [3 to 4]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 23 [6 to 92] | 11 [6 to 22] | 8 [5 to 14] | 14 [4 to 44] | 5 [2 to 13] | 38 [22 to 65] | 6 [3 to 12] | 53 [29 to 99] | 7 [4 to 13] | 16 [7 to 39] | 3 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GII.4: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run: Pre-Dose 1 | 21 [7 to 63] | 13 [5 to 34] | 5 [2 to 12] | 9 [4 to 20] | 23 [7 to 70] | 9 [3 to 29] | 5 [3 to 7] | 9 [4 to 23] | 6 [3 to 12] | 5 [2 to 9] | 6 [3 to 12]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 140 [92 to 213] | 193 [87 to 432] | 57 [24 to 138] | 52 [35 to 78] | 18 [6 to 53] | 92 [26 to 322] | 5 [3 to 8] | 41 [26 to 65] | 7 [3 to 14] | 96 [22 to 421] | 6 [3 to 13]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 120 [95 to 151] | 113 [53 to 239] | 27 [8 to 93] | 25 [14 to 42] | 16 [6 to 45] | 63 [21 to 186] | 5 [3 to 9] | 25 [9 to 70] | 7 [3 to 16] | 55 [18 to 170] | 6 [3 to 13]
  GII.4: I Run:28 Days PD1 | 116 [84 to 161] | 68 [32 to 149] | 19 [6 to 61] | 19 [10 to 34] | 19 [7 to 48] | 42 [11 to 159] | 5 [3 to 7] | 22 [9 to 55] | 6 [3 to 12] | 39 [15 to 100] | 6 [3 to 12]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 108 [73 to 160] | 94 [44 to 202] | 17 [6 to 48] | 22 [10 to 50] | 29 [12 to 72] | 44 [12 to 159] | 5 [3 to 8] | 22 [9 to 55] | 7 [3 to 14] | 36 [15 to 89] | 6 [3 to 11]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 108 [79 to 149] | 76 [36 to 174] | 19 [7 to 54] | 19 [9 to 39] | 30 [12 to 76] | 34 [10 to 117] | 5 [3 to 7] | 21 [9 to 53] | 6 [3 to 14] | 31 [13 to 73] | 6 [3 to 13]
  GII.4: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:Pre-Dose 1 | 8 [4 to 17] | 4 [2 to 7] | 4 [2 to 11] | 8 [4 to 17] | 5 [2 to 10] | 9 [3 to 28] | 5 [3 to 8] | 18 [5 to 66] | 8 [4 to 17] | 5 [2 to 12] | 7 [3 to 16]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 39 [22 to 71] | 32 [17 to 60] | 17 [7 to 42] | 19 [12 to 31] | 7 [3 to 20] | 38 [11 to 125] | 5 [3 to 9] | 44 [13 to 144] | 8 [4 to 19] | 42 [20 to 89] | 7 [3 to 16]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 25 [11 to 54] | 20 [9 to 44] | 9 [4 to 23] | 14 [7 to 28] | 6 [3 to 15] | 27 [9 to 83] | 6 [3 to 11] | 29 [10 to 85] | 9 [4 to 19] | 25 [10 to 65] | 6 [3 to 13]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 16 [5 to 45] | 13 [5 to 38] | 8 [3 to 22] | 16 [9 to 29] | 6 [3 to 11] | 17 [5 to 56] | 7 [3 to 18] | 24 [9 to 66] | 11 [4 to 28] | 19 [7 to 47] | 6 [3 to 13]

10. Secondary Outcome: GMT of Serum Anti-norovirus GI.1 and GII.4 VLP IgG
Description: as for outcome 9
Time Frame: I run: predose 1 and 7, 21, 28 days PD1, and 7 and 28 days PD2; II run: predose 1 and 28, 152 and 365 days PD2 (up to Day 393)
Population: PP population included all participants who received both doses of study product and with no protocol deviations likely to affect the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 9 | 9 | 8 | 7
titer
  GI.1: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run: Pre-Dose 1 | 13 [3 to 55] | 8 [2 to 27] | 28 [11 to 73] | 22 [7 to 68] | 9 [2 to 37] | 9 [3 to 26] | 7 [3 to 21] | 14 [5 to 38] | 11 [4 to 26] | 7 [2 to 32] | 5 [1 to 14]
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 211 [98 to 452] | 237 [120 to 466] | 1650 [673 to 4047] | 1171 [251 to 5457] | 5 [1 to 20] | 375 [97 to 1447] | 7 [2 to 19] | 96 [32 to 289] | 10 [4 to 24] | 82 [18 to 373] | 5 [1 to 16]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 266 [130 to 545] | 184 [93 to 363] | 1165 [495 to 2741] | 1235 [534 to 2858] | 7 [2 to 26] | 457 [159 to 1312] | 5 [1 to 18] | 97 [30 to 309] | 13 [5 to 30] | 107 [24 to 468] | 5 [1 to 14]
  GI.1: I Run:28 Days PD1 | 261 [140 to 486] | 152 [76 to 305] | 910 [379 to 2185] | 878 [409 to 1882] | 7 [2 to 26] | 429 [178 to 1036] | 6 [2 to 18] | 110 [41 to 300] | 10 [4 to 23] | 93 [22 to 395] | 5 [2 to 16]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 281 [152 to 520] | 167 [77 to 365] | 723 [360 to 1452] | 957 [554 to 1651] | 10 [2 to 49] | 513 [249 to 1060] | 7 [3 to 21] | 157 [66 to 373] | 10 [4 to 24] | 108 [25 to 474] | 5 [2 to 14]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 286 [151 to 540] | 168 [76 to 346] | 605 [256 to 1432] | 737 [399 to 1361] | 11 [2 to 50] | 518 [278 to 966] | 6 [2 to 19] | 177 [78 to 399] | 10 [4 to 26] | 127 [27 to 586] | 5 [2 to 16]
  GI.1: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:Pre-Dose 1 | 5 [2 to 14] | 7 [3 to 14] | 5 [3 to 8] | 5 [2 to 10] | 7 [2 to 27] | 8 [4 to 19] | 7 [3 to 14] | 9 [3 to 30] | 8 [4 to 18] | 3 [1 to 6] | 3 [1 to 5]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 83 [45 to 156] | 94 [46 to 192] | 89 [44 to 181] | 113 [78 to 164] | 10 [3 to 36] | 270 [178 to 411] | 6 [2 to 14] | 103 [53 to 200] | 8 [4 to 17] | 80 [56 to 116] | 3 [1 to 6]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 44 [22 to 91] | 65 [43 to 99] | 46 [24 to 89] | 73 [45 to 118] | 8 [2 to 28] | 135 [90 to 202] | 7 [3 to 16] | 82 [47 to 143] | 8 [4 to 17] | 35 [27 to 44] | 3 [1 to 5]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 58 [26 to 131] | 53 [40 to 68] | 28 [15 to 54] | 46 [23 to 92] | 6 [2 to 19] | 75 [55 to 103] | 6 [2 to 16] | 57 [33 to 99] | 10 [4 to 28] | 21 [13 to 34] | 3 [1 to 6]
  GII.4: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run: Pre-Dose 1 | 38 [10 to 142] | 19 [6 to 62] | 5 [2 to 14] | 17 [7 to 41] | 19 [5 to 69] | 8 [2 to 29] | 5 [2 to 15] | 10 [4 to 28] | 6 [2 to 20] | 11 [5 to 22] | 13 [4 to 45]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 97 [56 to 167] | 136 [66 to 279] | 43 [30 to 62] | 40 [27 to 60] | 14 [4 to 53] | 54 [14 to 206] | 5 [2 to 15] | 23 [14 to 37] | 9 [3 to 24] | 178 [100 to 317] | 16 [6 to 46]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 142 [70 to 286] | 128 [59 to 279] | 35 [25 to 50] | 39 [27 to 55] | 13 [4 to 45] | 93 [33 to 262] | 5 [2 to 15] | 29 [17 to 49] | 9 [3 to 28] | 180 [126 to 259] | 17 [6 to 48]
  GII.4: I Run:28 Days PD1 | 139 [73 to 267] | 98 [42 to 225] | 31 [22 to 45] | 37 [28 to 49] | 16 [6 to 46] | 86 [31 to 237] | 5 [2 to 13] | 30 [20 to 45] | 7 [2 to 20] | 148 [105 to 208] | 16 [6 to 45]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 144 [72 to 288] | 132 [71 to 248] | 34 [28 to 42] | 42 [34 to 51] | 25 [9 to 69] | 99 [42 to 233] | 5 [2 to 14] | 34 [25 to 45] | 8 [3 to 24] | 144 [106 to 196] | 15 [5 to 46]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 174 [90 to 336] | 125 [72 to 218] | 34 [26 to 46] | 41 [32 to 51] | 27 [10 to 75] | 102 [43 to 242] | 6 [2 to 15] | 36 [28 to 47] | 7 [3 to 21] | 140 [97 to 202] | 17 [6 to 49]
  GII.4: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:Pre-Dose 1 | 13 [5 to 31] | 11 [4 to 32] | 5 [2 to 13] | 10 [3 to 33] | 5 [2 to 14] | 6 [2 to 18] | 4 [2 to 9] | 9 [2 to 42] | 7 [2 to 20] | 3 [1 to 7] | 6 [2 to 14]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 65 [39 to 106] | 74 [46 to 120] | 57 [35 to 91] | 37 [18 to 73] | 8 [2 to 34] | 104 [65 to 166] | 5 [2 to 12] | 52 [22 to 120] | 7 [2 to 18] | 37 [25 to 56] | 6 [2 to 15]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 52 [31 to 87] | 44 [22 to 91] | 18 [8 to 41] | 18 [9 to 36] | 7 [2 to 23] | 77 [30 to 194] | 5 [2 to 11] | 33 [14 to 75] | 8 [2 to 26] | 20 [12 to 33] | 5 [2 to 12]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 28 [11 to 75] | 51 [27 to 96] | 13 [7 to 25] | 23 [11 to 51] | 6 [2 to 16] | 44 [24 to 81] | 6 [2 to 16] | 22 [9 to 54] | 13 [5 to 34] | 16 [8 to 34] | 5 [2 to 12]

11. Secondary Outcome: GMT of Serum Anti-norovirus GI.1 and GII.4 VLP IgM
Description: as for outcome 9
Time Frame: as for outcome 10
Population: Data was not collected because serum specimens were not tested for specific IgM antibodies to Norovirus GI.1 and GII.4 VLPs as per the change in planned analysis, because this measurement was not informative in a previous study LV01-103 (NCT00973284).
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Serum Anti-norovirus GI.1 and GII.4 VLP IgA as Compared to Baseline
Description: as for outcome 9
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: PP population where baseline and specified post-baseline assessment were available. PP population included all participants who received both doses of study product and with no protocol deviations likely to affect the immunogenicity assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
fold rise
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 23.1 [7.4 to 71.9] | 76.1 [38.1 to 152] | 84.4 [20.6 to 345.1] | 122.9 [30 to 503.7] | 0.8 [0.3 to 1.8] | 115.2 [35.5 to 373.7] | 1 [1 to 1] | 39.1 [10.3 to 148.2] | 1 [1 to 1] | 12.6 [4.2 to 37.6] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 18.5 [7 to 49] | 34.9 [16.6 to 73.4] | 49.6 [18.2 to 134.9] | 52.1 [19.3 to 140.4] | 1 [0.9 to 1.2] | 81.2 [48.6 to 135.7] | 1 [0.9 to 1.1] | 24.2 [6.9 to 85.7] | 1 [0.9 to 1] | 9.7 [3.1 to 30.2] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:28 Days PD1 | 16.2 [6.1 to 42.8] | 22.6 [11.1 to 46] | 33.7 [11.7 to 46] | 25.4 [10.5 to 61.3] | 1 [0.8 to 1.2] | 57.5 [30.6 to 108] | 1 [0.9 to 1.1] | 19.6 [6.4 to 60.5] | 1 [0.9 to 1] | 6.6 [2.4 to 18.8] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 15.1 [6.2 to 37] | 22.5 [11.8 to 42.9] | 23.9 [9.6 to 59.7] | 22.2 [10.8 to 45.4] | 1.1 [0.7 to 1.6] | 45.2 [23.4 to 87.2] | 1 [1 to 1.1] | 19.7 [7.3 to 53.2] | 1 [0.9 to 1] | 6 [2.1 to 17.3] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 13 [5 to 33.6] | 16 [7.4 to 34.5] | 12.1 [4.8 to 30.7] | 13.2 [5 to 34.7] | 1 [0.7 to 1.3] | 31.3 [15.4 to 63.7] | 1.1 [0.9 to 1.3] | 14.2 [5.1 to 39.8] | 1 [1 to 1.1] | 5.3 [2.1 to 13.1] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 7 [3.7 to 13.3] | 5 [2.3 to 10.7] | 3.6 [1.9 to 6.8] | 4.7 [1.9 to 11.7] | 1 [1 to 1] | 38.6 [19.9 to 74.6] | 1 [0.9 to 1.1] | 25.5 [9.1 to 71.4] | 1 [1 to 1] | 9.6 [3.7 to 24.9] | 1.1 [0.9 to 1.5]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 3.6 [1.8 to 7.1] | 4.1 [2 to 8.3] | 3.3 [1.8 to 6] | 4.6 [1.7 to 12] | 1 [1 to 1] | 18.5 [11.5 to 29.8] | 1.1 [0.9 to 1.3] | 12.9 [5.5 to 30] | 1.1 [0.9 to 1.3] | 6.6 [2.9 to 15.1] | 1.1 [0.9 to 1.4]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 4.1 [1.3 to 13.5] | 3.7 [1.9 to 7.1] | 2.6 [1.6 to 4.4] | 4.5 [1.4 to 14.1] | 1 [0.9 to 1] | 12.2 [7.1 to 20.9] | 1 [0.9 to 1.2] | 8.8 [3.9 to 20.2] | 1.3 [0.9 to 1.9] | 5.2 [2.1 to 12.7] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data.
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 6.7 [2.2 to 20.7] | 15.4 [4.7 to 50.8] | 10.7 [3.5 to 32.9] | 5 [2.2 to 11] | 1 [0.9 to 1.1] | 9.7 [3 to 30.6] | 1 [1 to 1.1] | 4.4 [2.1 to 9.6] | 1.2 [0.9 to 1.4] | 19.9 [5.9 to 67.6] | 1 [1 to 1.1]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 5.7 [2 to 16.5] | 9 [4.1 to 20] | 5 [1.3 to 18.9] | 2.7 [1.3 to 5.5] | 0.9 [0.7 to 1] | 6.6 [3 to 14.4] | 1.1 [0.9 to 1.2] | 3.5 [1.2 to 9.7] | 1.1 [0.8 to 1.6] | 11.4 [3.9 to 33.3] | 1 [1 to 1.1]
  GII.4: I Run:28 Days PD1 | 5.6 [2.1 to 14.8] | 5.5 [2.4 to 12.3] | 3.6 [1.1 to 12] | 2 [1 to 4.3] | 1 [0.6 to 1.9] | 4.5 [1.9 to 10.7] | 1 [0.9 to 1.1] | 2.4 [0.9 to 6.4] | 1 [0.8 to 1.2] | 8.1 [3.2 to 20.4] | 1 [0.9 to 1.1]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 5.2 [2.1 to 12.6] | 6.1 [2.9 to 12.7] | 3.2 [1.1 to 9.4] | 2.5 [1 to 5.9] | 1.3 [0.4 to 3.6] | 4.6 [2.1 to 10.3] | 1.1 [1 to 1.1] | 2.4 [0.9 to 6.3] | 1.1 [0.9 to 1.5] | 7.5 [3 to 18.6] | 1 [0.8 to 1.1]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 5.2 [2.1 to 12.6] | 5.2 [2.6 to 10.2] | 3.4 [1.4 to 8.4] | 2 [1 to 4.4] | 1.3 [0.5 to 3.3] | 3.5 [1.7 to 7.4] | 1 [1 to 1.1] | 2.3 [1 to 5.7] | 1.1 [0.9 to 1.4] | 6.4 [2.6 to 15.6] | 1.1 [1 to 1.2]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 4.7 [2.9 to 7.7] | 7.5 [4.6 to 12.2] | 3.9 [1.6 to 9.1] | 2.5 [1 to 5.9] | 1.5 [0.6 to 3.6] | 4 [1.9 to 8.3] | 1.1 [0.9 to 1.4] | 2.4 [0.8 to 7.2] | 1 [0.9 to 1.2] | 8.1 [3.2 to 20.4] | 1 [0.9 to 1]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 2.6 [1.8 to 3.9] | 4.8 [2.4 to 9.4] | 2 [1 to 4] | 1.9 [0.8 to 4.5] | 1.3 [0.7 to 2.4] | 2.8 [1.5 to 5.2] | 1.2 [0.9 to 1.6] | 1.6 [0.5 to 4.8] | 1.1 [0.9 to 1.4] | 4.8 [1.8 to 12.7] | 0.8 [0.6 to 1.2]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 2 [1.2 to 3.2] | 3.1 [1.3 to 7.3] | 1.7 [0.9 to 3.5] | 1.8 [0.8 to 4.2] | 1.3 [0.8 to 2.1] | 1.8 [0.9 to 3.6] | 1.5 [0.9 to 2.6] | 1.3 [0.4 to 4.1] | 1.4 [0.8 to 2.3] | 4.4 [1.6 to 12] | 0.8 [0.6 to 1.1]

13. Secondary Outcome: GMFR of Serum Anti-norovirus GI.1 and GII.4 VLP IgG as Compared to Baseline
Description: as for outcome 9
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
fold rise
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 16.2 [3.8 to 68.7] | 29.4 [11.2 to 77.2] | 59.5 [27.2 to 130.2] | 54.9 [17.6 to 171] | 0.7 [0.2 to 2] | 43 [5.9 to 315.7] | 0.9 [0.6 to 1.4] | 6.8 [2.3 to 20.8] | 0.9 [0.8 to 1] | 11.2 [2.4 to 52.4] | 1 [0.9 to 1.1]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 20.5 [5.2 to 80.2] | 22.8 [8.7 to 59.8] | 42 [22.6 to 78.3] | 55.2 [25.7 to 118.7] | 1 [0.8 to 1.2] | 52.5 [10.2 to 270.8] | 0.8 [0.5 to 1.2] | 7.5 [2.4 to 23.1] | 0.9 [0.8 to 1.1] | 14.4 [2.9 to 71.8] | 1 [0.9 to 1.1]
  GI.1: I Run:28 Days PD1 | 20 [4.9 to 81.6] | 18.9 [6.8 to 52.6] | 32.8 [18.2 to 59.2] | 39.2 [17.6 to 87.6] | 1 [0.8 to 1.2] | 49.3 [11.2 to 217.8] | 0.8 [0.5 to 1.3] | 7.9 [3.1 to 20.4] | 0.9 [0.8 to 1] | 12.7 [2.7 to 59.3] | 1.1 [0.9 to 1.2]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 21.6 [5.4 to 86.1] | 23.8 [9 to 63.2] | 26.1 [15.2 to 44.8] | 42.8 [17.4 to 104.8] | 1.2 [0.7 to 2.1] | 59 [14.4 to 241] | 1 [0.6 to 1.7] | 11.3 [4.3 to 29.8] | 0.9 [0.8 to 1] | 14.7 [3.1 to 70.3] | 1 [0.8 to 1.2]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 22 [5.6 to 86.3] | 23.1 [8.8 to 60.6] | 19.7 [11.8 to 32.9] | 32.9 [14.6 to 74.5] | 1.2 [0.8 to 1.9] | 59.5 [16.9 to 209.6] | 0.9 [0.5 to 1.5] | 12.6 [4.9 to 32.8] | 0.9 [0.9 to 1] | 17.2 [3.6 to 82.7] | 1.1 [0.9 to 1.2]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 17 [4.9 to 59.2] | 14.1 [7.9 to 25.3] | 18.8 [9.3 to 37.9] | 23.9 [14.4 to 39.7] | 1.4 [0.8 to 2.5] | 32 [14.5 to 70.5] | 0.8 [0.6 to 1.3] | 10.9 [3.8 to 31] | 1 [0.8 to 1.2] | 26.6 [11.2 to 63] | 1.1 [0.9 to 1.3]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 7.9 [2.3 to 26.6] | 9.8 [5.2 to 18.5] | 9.6 [5.1 to 18] | 15.5 [7.1 to 33.9] | 1.1 [0.7 to 1.9] | 15.9 [6.5 to 38.9] | 1 [0.7 to 1.4] | 8.7 [3.3 to 22.7] | 1 [0.7 to 1.3] | 11.5 [5.1 to 26] | 0.9 [0.6 to 1.3]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 9.3 [1.7 to 49.5] | 7.9 [4.1 to 14.9] | 6.1 [3.6 to 10.4] | 11.7 [5 to 27.4] | 1.1 [0.6 to 2.1] | 8.9 [4.1 to 19.3] | 0.9 [0.5 to 1.6] | 6 [2.4 to 15] | 1.3 [0.7 to 2.5] | 8.2 [3.6 to 18.6] | 1 [0.9 to 1.2]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 2.6 [0.8 to 8.3] | 7.1 [2.4 to 20.3] | 8.3 [3.4 to 20.1] | 2.4 [1.1 to 5.1] | 1 [0.9 to 1.1] | 6.8 [2.2 to 21.1] | 1 [1 to 1.1] | 2.3 [1.2 to 4.4] | 1.4 [0.9 to 2] | 16.1 [5.7 to 45.4] | 1.3 [1 to 1.6]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 3.8 [1.1 to 12.8] | 6.6 [2.5 to 17.6] | 6.8 [2.8 to 16.1] | 2.3 [1.2 to 4.2] | 0.9 [0.8 to 1] | 11.7 [4.7 to 29.2] | 1 [0.9 to 1.1] | 3.3 [1.4 to 8] | 1.3 [0.9 to 1.8] | 16.4 [7 to 38.3] | 1.4 [1 to 1.8]
  GII.4: I Run:28 Days PD1 | 3.7 [1.1 to 12.8] | 5.1 [1.9 to 13.4] | 6 [2.6 to 14.3] | 2.2 [1.1 to 4.4] | 1.1 [0.6 to 2.2] | 10.8 [4.2 to 27.9] | 0.9 [0.9 to 1] | 3 [1.4 to 6.4] | 1 [0.9 to 1.2] | 13.4 [5.7 to 31.6] | 1.3 [1 to 1.6]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 3.8 [1.1 to 13.9] | 4.8 [1.8 to 12.6] | 6.6 [2.7 to 16.1] | 2.5 [1.1 to 5.5] | 1.4 [0.5 to 4.1] | 12.3 [4.6 to 32.6] | 1 [0.9 to 1.1] | 3.4 [1.4 to 7.9] | 1.2 [1 to 1.6] | 13.1 [6.1 to 27.8] | 1.2 [0.9 to 1.5]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 4.6 [1.3 to 16.3] | 4.6 [1.8 to 11.6] | 5.8 [2.5 to 13.8] | 2.4 [1.2 to 5] | 1.5 [0.5 to 4.5] | 12.8 [4.6 to 35.5] | 1.1 [0.9 to 1.3] | 3.7 [1.6 to 8.5] | 1.1 [0.9 to 1.4] | 12.7 [6.3 to 25.5] | 1.3 [1 to 1.8]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 5 [2.3 to 10.8] | 6.8 [2.8 to 16.4] | 12 [5.5 to 26.2] | 3.5 [1.1 to 11.5] | 1.6 [0.5 to 4.5] | 18.1 [4.4 to 74.6] | 1.3 [1 to 1.6] | 5.7 [1.7 to 19.6] | 1 [0.7 to 1.5] | 12.2 [5.7 to 26.3] | 1 [0.9 to 1.2]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 3.1 [1.4 to 6.7] | 4 [1.6 to 10] | 3.9 [1.5 to 10] | 1.7 [0.7 to 4.2] | 1.4 [0.8 to 2.6] | 13.4 [3.4 to 51.9] | 1.2 [0.8 to 1.8] | 3.6 [0.9 to 14.9] | 1.2 [0.6 to 2.3] | 6.5 [3.4 to 12.2] | 0.9 [0.6 to 1.2]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 2.7 [1 to 7.4] | 4.6 [2 to 10.6] | 2.4 [0.8 to 7.5] | 1.9 [0.6 to 5.9] | 1.3 [0.7 to 2.5] | 7.7 [2.5 to 23.7] | 1.4 [0.8 to 2.5] | 2.5 [0.6 to 9.9] | 1.9 [0.9 to 4.3] | 6 [3.2 to 11.2] | 0.9 [0.7 to 1.1]

14. Secondary Outcome: GMFR of Serum Anti-norovirus GI.1 and GII.4 VLP IgM as Compared to Baseline
Description: as for outcome 9
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 11
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants With Seroresponse for Serum Anti-norovirus GI.1 and GII.4 VLP IgA
Description: Seroresponse was defined as a 4-fold increase in antibody titer compared to pre-immunization titers. Run I was defined as the initial analysis performed once Day 56 post dose data was available. Run II was defined as final analysis performed after all later time points were achieved.
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
percentage of participants
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 77.8 [40.0 to 97.2] | 100.0 [63.1 to 100.0] | 90.0 [55.5 to 99.7] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 88.9 [51.8 to 99.7] | 100.0 [63.1 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 36.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD1 | 77.8 [40.0 to 97.2] | 100.0 [63.1 to 100.0] | 90.0 [55.5 to 99.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 88.9 [51.8 to 99.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 66.7 [29.9 to 92.5] | 71.4 [29.0 to 96.3] | 55.6 [21.2 to 86.3] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 100.0 [66.4 to 100.0] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 62.5 [24.5 to 91.5] | 42.9 [9.9 to 81.6] | 44.4 [13.7 to 78.8] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 41.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 50.0 [11.8 to 88.2] | 42.9 [9.9 to 81.6] | 37.5 [8.5 to 75.5] | 57.1 [18.4 to 90.1] | 0.0 [0.0 to 41.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 33.6] | 71.4 [29.0 to 96.3] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 55.6 [21.2 to 86.3] | 75.0 [34.9 to 96.8] | 70.0 [34.8 to 93.3] | 42.9 [9.9 to 81.6] | 0.0 [0.0 to 36.9] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 30.8] | 55.6 [21.2 to 86.3] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 55.6 [21.2 to 86.3] | 75.0 [34.9 to 96.8] | 50.0 [18.7 to 81.3] | 25.0 [3.2 to 65.1] | 0.0 [0.0 to 36.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 30.8] | 25.0 [3.2 to 65.1] | 0.0 [0.0 to 36.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD1 | 55.6 [21.2 to 86.3] | 62.5 [24.5 to 91.5] | 50.0 [18.7 to 81.3] | 12.5 [0.3 to 52.7] | 12.5 [0.3 to 52.7] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 30.8] | 22.2 [2.8 to 60.0] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 44.4 [13.7 to 78.8] | 71.4 [29.0 to 96.3] | 50.0 [18.7 to 81.3] | 25.0 [3.2 to 65.1] | 12.5 [0.3 to 52.7] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 30.8] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 44.4 [13.7 to 78.8] | 57.1 [18.4 to 90.1] | 44.4 [13.7 to 78.8] | 25.0 [3.2 to 65.1] | 12.5 [0.3 to 52.7] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 30.8] | 22.2 [2.8 to 60.0] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 55.6 [21.2 to 86.3] | 37.5 [8.5 to 75.5] | 14.3 [0.4 to 57.9] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 30.8] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 33.6] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 41.0]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 12.5 [0.3 to 52.7] | 42.9 [9.9 to 81.6] | 33.3 [7.5 to 70.1] | 25.0 [3.2 to 65.1] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1] | 0.0 [0.0 to 30.8] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 33.6] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 41.0]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 0.0 [0.0 to 45.9] | 42.6 [9.9 to 81.6] | 37.5 [8.5 to 75.5] | 14.3 [0.4 to 57.9] | 14.3 [0.4 to 57.9] | 25.0 [3.2 to 65.1] | 10.0 [0.3 to 44.5] | 22.2 [2.8 to 60.0] | 11.1 [0.3 to 48.2] | 57.1 [18.4 to 90.1] | 0.0 [0.0 to 41.0]

16. Secondary Outcome: Percentage of Participants With Seroresponse for Serum Anti-norovirus GI.1 and GII.4 VLP IgG
Description: as for outcome 15
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
percentage of participants
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 66.7 [29.9 to 92.5] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 55.6 [21.2 to 86.3] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 9 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 77.8 [40.0 to 97.2] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 33.6] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 36.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD1 | 77.8 [40.0 to 97.2] | 87.5 [47.3 to 99.7] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 55.6 [21.2 to 86.3] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 12.5 [0.3 to 52.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 12.5 [0.3 to 52.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 77.8 [40.0 to 97.2] | 100.0 [59.0 to 100.0] | 88.9 [51.8 to 99.7] | 100.0 [63.1 to 100.0] | 14.3 [0.4 to 57.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 50.0 [15.7 to 84.3] | 85.7 [42.1 to 99.6] | 88.9 [51.8 to 99.7] | 87.5 [47.3 to 99.7] | 14.3 [0.4 to 57.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 50.0 [11.8 to 88.2] | 85.7 [42.1 to 99.6] | 75.0 [34.9 to 96.8] | 85.7 [42.1 to 99.6] | 0.0 [0.0 to 41.0] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 11.1 [0.3 to 48.2] | 71.4 [29.0 to 96.3] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 22.2 [2.8 to 60.0] | 62.5 [24.5 to 91.5] | 80.0 [44.4 to 97.5] | 28.6 [3.7 to 871.0] | 0.0 [0.0 to 36.9] | 62.5 [24.5 to 91.5] | 0.0 [0.0 to 30.8] | 33.3 [7.5 to 70.1] | 0.0 [0.0 to 33.6] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 33.3 [7.5 to 70.1] | 62.5 [24.5 to 91.5] | 70.0 [34.8 to 93.3] | 12.5 [0.3 to 52.7] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 50.0 [15.7 to 84.3] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD1 | 33.3 [7.5 to 70.1] | 62.5 [24.5 to 91.5] | 70.0 [34.8 to 93.3] | 12.5 [0.3 to 52.7] | 12.5 [0.3 to 52.7] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 30.8] | 44.4 [13.7 to 878.8] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 44.4 [13.7 to 78.8] | 57.1 [18.4 to 90.1] | 70.0 [34.8 to 93.3] | 25.0 [3.2 to 65.1] | 12.5 [0.3 to 52.7] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 30.8] | 44.4 [13.7 to 78.8] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 33.3 [7.5 to 70.1] | 57.1 [18.4 to 90.1] | 66.7 [29.9 to 92.5] | 12.5 [0.3 to 52.7] | 12.5 [0.3 to 52.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 44.4 [13.7 to 78.8] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 55.6 [21.2 to 86.3] | 71.4 [29.0 to 96.3] | 77.8 [40.0 to 97.2] | 50.0 [15.7 to 84.3] | 14.3 [0.4 to 57.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 50.0 [15.7 to 84.3] | 42.9 [9.9 to 81.6] | 66.7 [29.9 to 92.5] | 25.0 [3.5 to 65.1] | 14.3 [0.4 to 57.9] | 62.5 [24.5 to 91.5] | 10.0 [0.3 to 44.5] | 66.7 [29.9 to 92.5] | 11.1 [0.3 to 48.2] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 41.0]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 33.3 [4.3 to 77.7] | 57.1 [18.4 to 90.1] | 50.0 [15.7 to 584.3] | 28.6 [3.7 to 71.0] | 14.3 [0.4 to 57.9] | 50.0 [15.7 to 84.3] | 10.0 [0.3 to 44.5] | 55.6 [21.2 to 86.3] | 22.2 [2.8 to 60.0] | 85.7 [42.1 to 99.6] | 0.0 [0.0 to 41.0]

17. Secondary Outcome: Percentage of Participants With Seroresponse for Serum Anti-norovirus GI.1 and GII.4 VLP IgM
Description: as for outcome 15
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 11
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: GMT of Anti-norovirus GI.1 and GII.4 VLP IgA, IgG, and IgM Combined Using Pan-Ig Enzyme-Linked Immunosorbent Assay (ELISA)
Description: GMTs were assessed for Anti-norovirus GI.1 and GII.4 VLP by Pan-Ig ELISA. A pan ELISA assay captured IgG, IgA and IgM combined. Run I was defined as the initial analysis performed once Day 56 post dose data was available. Run II was defined as final analysis performed after all later time points were achieved.
Time Frame: I run: predose 1, 7, 21, 28 days PD1, 7 and 28 days PD2; II run: predose 1, 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 9 | 9 | 8 | 7
titer
  GI.1: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run: Pre-Dose 1 | 3763 [894 to 15838] | 2348 [599 to 9198] | 2560 [950 to 6901] | 2153 [447 to 10366] | 1396 [162 to 12052] | 1810 [486 to 6737] | 2744 [806 to 9337] | 6451 [2020 to 20603] | 2763 [668 to 21197] | 1280 [320 to 5115] | 861 [147 to 5054]
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 163840 [77123 to 348063] | 231705 [135499 to 396217] | 351199 [159240 to 774559] | 220512 [57489 to 831259] | 1185 [179 to 7861] | 150242 [52704 to 428288] | 2229 [596 to 8327] | 151695 [57115 to 402894] | 3763 [668 to 21197] | 126338 [39749 to 401554] | 861 [153 to 4860]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 260080 [122425 to 552516] | 194840 [92705 to 409496] | 285262 [127800 to 636731] | 212474 [93970 to 480425] | 1185 [193 to 7282] | 212474 [114914 to 392862] | 2389 [658 to 8676] | 115852 [51050 to 262916] | 7241 [2719 to 19283] | 137772 [58166 to 326329] | 861 [207 to 3587]
  GI.1: I Run:28 Days PD1 | 222952 [109569 to 453664] | 126338 [59394 to 268734] | 216188 [102476 to 456081] | 194840 [106949 to 354959] | 1280 [219 to 7493] | 212474 [106756 to 422883] | 2389 [658 to 8676] | 120401 [56380 to 257117] | 3763 [696 to 20334] | 106230 [42084 to 268187] | 707 [122 to 4078]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 176957 [85545 to 366049] | 163840 [86301 to 311047] | 266159 [143088 to 495085] | 212474 [124953 to 361298] | 1974 [396 to 9852] | 231705 [169986 to 315832] | 2229 [584 to 8500] | 176957 [116676 to 268383] | 4389 [872 to 22081] | 126338 [68328 to 233597] | 861 [207 to 3587]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 206425 [102014 to 417702] | 148394 [83353 to 264185] | 176957 [81595 to 383771] | 150242 [92634 to 243676] | 1974 [352 to 11056] | 300484 [156475 to 577028] | 2079 [532 to 8134] | 176957 [128475 to 243735] | 5120 [1388 to 18883] | 89334 [61622 to 129510] | 861 [180 to 4116]
  GI.1: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:Pre-Dose 1 | 4389 [978 to 19405] | 3121 [657 to 14817] | 3484 [870 to 13946] | 1974 [408 to 9540] | 3121 [415 to 23466] | 2560 [803 to 8158] | 2941 [804 to 10760] | 4389 [156 to 12222] | 2560 [567 to 11554] | 587 [155 to 2219] | 390 [82 to 1852]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 260080 [112007 to 603906] | 243465 [117694 to 503640] | 222952 [91740 to 541832] | 212474 [124953 to 361298] | 3446 [506 to 23456] | 357338 [246486 to 518042] | 2744 [696 to 10819] | 140451 [98461 to 200348] | 2195 [392 to 12279] | 89334 [61622 to 129510] | 353 [53 to 2369]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 97420 [41130 to 230749] | 121733 [53847 to 275205] | 95562 [43402 to 210408] | 126338 [93602 to 170523] | 3121 [478 to 20386] | 150242 [103635 to 217810] | 2941 [756 to 11445] | 81920 [56204 to 119401] | 2370 [409 to 13721] | 31584 [20522 to 48609] | 390 [75 to 2018]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 145965 [62364 to 341636] | 67202 [25756 to 175341] | 63169 [21663 to 184198] | 81920 [48537 to 138264] | 2153 [409 to 11331] | 75121 [51817 to 108905] | 2941 [699 to 12376] | 47781 [30650 to 74487] | 3484 [560 to 21684] | 18549 [10419 to 33023] | 353 [64 to 1960]
  GII.4: I Run: Pre-Dose 1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run: Pre-Dose 1 | 11945 [3089 to 46196] | 3948 [1103 to 14126] | 1470 [287 to 7526] | 28963 [5792 to 144824] | 5583 [1425 to 21877] | 4695 [804 to 27403] | 2229 [408 to 12181] | 9481 [1706 to 52683] | 8127 [1540 to 42902] | 6089 [2015 to 18402] | 9275 [2069 to 41572]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 9 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 55738 [32476 to 95661] | 53119 [23492 to 120106] | 71316 [35649 to 142667] | 593575 [250592 to 1405995] | 4740 [1381 to 16278] | 115852 [45745 to 293407] | 1940 [377 to 9997] | 88478 [42773 to 183024] | 6451 [1429 to 29113] | 300484 [110464 to 817377] | 7608 [1665 to 34773]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 9 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 70225 [39229 to 125714] | 44667 [20355 to 98017] | 50428 [24962 to 101872] | 505352 [297190 to 859315] | 5120 [1603 to 16352] | 163840 [81963 to 327507] | 1810 [329 to 9966] | 126338 [55875 to 285662] | 9390 [1854 to 47567] | 212474 [114914 to 392862] | 8400 [1694 to 41653]
  GII.4: I Run:28 Days PD1 | 70225 [33407 to 147623] | 40960 [19180 to 87472] | 38217 [17951 to 81361] | 275545 [151249 to 501988] | 6451 [2151 to 19348] | 150242 [84602 to 266810] | 2079 [426 to 10158] | 111476 [52201 to 238058] | 7525 [1588 to 35664] | 126338 [74298 to 214829] | 7608 [1665 to 34773]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 75848 [40737 to 141221] | 60866 [36756 to 100792] | 43900 [24247 to 79483] | 300484 [185267 to 487353] | 10240 [3502 to 29943] | 163840 [88181 to 304413] | 1810 [329 to 9966] | 130040 [67714 to 249731] | 8127 [1573 to 41991] | 178669 [100609 to 317292] | 10240 [2130 to 49233]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 75848 [34973 to 164493] | 60866 [36756 to 100792] | 47781 [25186 to 90647] | 212474 [106756 to 422883] | 11167 [3442 to 36230] | 126338 [68328 to 233597] | 1810 [363 to 9026] | 103213 [46414 to 229521] | 6967 [1405 to 34539] | 115852 [57957 to 231582] | 10240 [2330 to 45004]
  GII.4: II Run:Pre-Dose 1: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:Pre-Dose 1 | 13934 [3481 to 55783] | 10240 [2841 to 36907] | 4389 [1026 to 18781] | 18780 [3498 to 100825] | 4200 [968 to 18216] | 3948 [544 to 28648] | 2560 [606 to 10815] | 7525 [1257 to 45038] | 6967 [1540 to 31526] | 5120 [2022 to 12967] | 5653 [1106 to 28892]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 88478 [44992 to 173997] | 90447 [38184 to 214241] | 103213 [65064 to 163729] | 126338 [63477 to 251448] | 8400 [1240 to 56896] | 150242 [78238 to 288514] | 2560 [727 to 9014] | 65020 [32132 to 131568] | 6967 [1577 to 30788] | 115852 [62354 to 215253] | 6241 [1439 to 27068]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 81920 [34112 to 196732] | 49931 [24467 to 101894] | 27869 [15260 to 50896] | 63169 [34164 to 116798] | 6241 [1158 to 33639] | 150242 [48269 to 467639] | 2744 [740 to 10177] | 35113 [14643 to 84196] | 8778 [2002 to 38482] | 48710 [23176 to 102374] | 5653 [1321 to 24190]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 8 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 45976 [13134 to 160938] | 49931 [19137 to 130278] | 20480 [11977 to 35021] | 67202 [25756 to 175341] | 3948 [957 to 16290] | 57926 [33875 to 99054] | 3378 [690 to 16544] | 27869 [11467 to 67729] | 12902 [3151 to 52826] | 37098 [17025 to 80838] | 5653 [1321 to 24190]

19. Secondary Outcome: GMFR of Anti-norovirus GI.1 and GII.4 VLP IgA, IgG, and IgM Combined Using Pan-Ig ELISA as Compared to Baseline
Description: GMFRs in GMTs of Anti-norovirus GI.1 and GII.4 VLP by Pan-Ig ELISA. A pan ELISA assay captured IgG, IgA and IgM combined. Run I was defined as the initial analysis performed once Day 56 post dose data was available. Run II was defined as final analysis performed after all later time points were achieved.
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
fold rise
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 43.5 [9.9 to 192.4] | 98.7 [21.7 to 449.2] | 137.2 [50.3 to 374.4] | 128 [61.1 to 268.3] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 83 [9.7 to 708.7] | 0.8 [0.6 to 1] | 23.5 [5.5 to 101.4] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 98.7 [28.7 to 339.9] | 1 [0.7 to 1.4]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 69.1 [15.9 to 300.6] | 83 [17.7 to 389.8] | 111.4 [51.7 to 240.2] | 98.7 [41.2 to 236.2] | 1.1 [0.8 to 1.6] | 117.4 [23.2 to 594.6] | 0.9 [0.7 to 1.1] | 20.7 [4.2 to 103.6] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 107.6 [23.8 to 487] | 1 [0.6 to 1.7]
  GI.1: I Run:28 Days PD1 | 59.3 [12.4 to 283] | 53.8 [11.5 to 251.3] | 84.4 [49.6 to 143.9] | 90.5 [31 to 264.7] | 1.2 [0.8 to 1.8] | 117.4 [19.1 to 722.8] | 0.9 [0.7 to 1.1] | 18.7 [5.7 to 61] | 1 [0.8 to 1.3] | 83 [18.2 to 377.8] | 0.8 [0.6 to 1.1]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 47 [8.9 to 248.9] | 78 [15.1 to 403.5] | 104 [58.5 to 184.8] | 98.7 [31.1 to 313.7] | 1.4 [0.6 to 3.2] | 128 [29 to 565.4] | 0.8 [0.6 to 1] | 27.4 [8.9 to 84.3] | 1.2 [0.9 to 1.5] | 98.7 [28.7 to 339.9] | 1 [0.6 to 1.7]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 54.9 [10.2 to 294.4] | 70.7 [16.5 to 302.4] | 64 [37.6 to 109] | 69.8 [20.7 to 235.7] | 1.4 [0.6 to 3.2] | 166 [35.3 to 779.6] | 0.8 [0.5 to 1.1] | 27.4 [9.9 to 76.4] | 1.4 [0.7 to 2.5] | 69.8 [19.9 to 245] | 1 [0.7 to 1.4]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 59.3 [13 to 270.2] | 78 [16.4 to 370.4] | 64 [31.6 to 129.5] | 107.6 [34.1 to 339.4] | 1.1 [0.6 to 2] | 139.6 [46.8 to 416.2] | 0.9 [0.6 to 1.3] | 32 [12.2 to 83.6] | 0.9 [0.7 to 1.1] | 152.2 [41.3 to 561.3] | 0.9 [0.6 to 1.4]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 17.4 [4.3 to 70.8] | 39 [7.9 to 193.4] | 27.4 [11.9 to 63.1] | 64 [15 to 273.6] | 1 [0.7 to 1.4] | 58.7 [21.6 to 159.6] | 1 [0.7 to 1.5] | 18.7 [8.5 to 41.1] | 0.9 [0.7 to 1.3] | 53.8 [15.7 to 184] | 1 [0.7 to 1.4]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 25.4 [2.1 to 311.2] | 21.5 [4.7 to 98.4] | 19 [8.5 to 42.5] | 58 [16.6 to 202.6] | 1 [0.6 to 1.7] | 29.3 [10.8 to 79.8] | 1 [0.7 to 1.5] | 10.9 [3.7 to 31.7] | 1.4 [0.7 to 2.5] | 43.1 [19.7 to 97.4] | 0.9 [0.6 to 1.4]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 4.7 [1.5 to 14.3] | 13.5 [3 to 60.9] | 48.5 [7.9 to 297.4] | 19.5 [1.8 to 213] | 1 [NA to NA] — Confidence interval could not be calculated because there was no variance in the observed data. | 24.7 [4.7 to 130.6] | 0.9 [0.6 to 1.2] | 9.3 [2.2 to 39.9] | 0.8 [0.6 to 1] | 49.4 [9.6 to 253.7] | 0.8 [0.6 to 1.1]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 5.9 [1.5 to 23.5] | 11.3 [3.6 to 36.1] | 34.3 [7.3 to 160.1] | 17.4 [3.2 to 96.4] | 1.1 [0.8 to 1.6] | 34.9 [7.1 to 171.6] | 0.8 [0.6 to 1.1] | 19 [5.4 to 67.6] | 0.8 [0.6 to 1.1] | 34.9 [7.5 to 131.4] | 0.9 [0.6 to 1.4]
  GII.4: I Run:28 Days PD1 | 5.9 [1.5 to 22.3] | 10.4 [3.6 to 30.3] | 26 [5.1 to 131.4] | 9.5 [1.8 to 50.1] | 1.4 [0.8 to 2.6] | 32 [7.7 to 132.3] | 0.9 [0.7 to 1.2] | 11.8 [3 to 45.9] | 0.9 [0.8 to 1.1] | 20.7 [5.2 to 82.7] | 0.8 [0.6 to 1.1]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 6.3 [2 to 20.3] | 10.8 [2.9 to 40.6] | 29.9 [6.1 to 146.9] | 10.4 [2.1 to 50.2] | 1.8 [0.5 to 6.2] | 34.9 [6.3 to 192.7] | 0.8 [0.6 to 1.1] | 13.7 [3.1 to 60.1] | 1 [0.8 to 1.3] | 29.3 [8.4 to 103] | 1.1 [0.7 to 1.7]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 6.3 [1.7 to 24.1] | 10.8 [3.4 to 34.4] | 21.8 [6.6 to 71.9] | 7.3 [1.5 to 35] | 2 [0.5 to 8.3] | 26.9 [5.4 to 133.6] | 0.8 [0.6 to 1.1] | 10.9 [2.5 to 48.1] | 0.9 [0.7 to 1.1] | 19 [5.4 to 67.6] | 1.1 [0.7 to 1.7]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 6.3 [1.6 to 24.7] | 8.8 [2.5 to 30.9] | 23.5 [6.5 to 84.6] | 6.7 [1.5 to 29.5] | 2 [0.5 to 8.4] | 38.1 [6 to 242.5] | 1 [0.8 to 1.3] | 8.6 [1.9 to 40.3] | 1 [0.8 to 1.3] | 22.6 [8.5 to 60.3] | 1.1 [0.9 to 1.4]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 3.7 [1.5 to 9] | 4.9 [1.4 to 17.3] | 6.3 [1.9 to 21.5] | 3.4 [0.8 to 13.3] | 1.5 [0.5 to 4.2] | 38.1 [7 to 206.1] | 1.1 [0.7 to 1.7] | 4.7 [0.9 to 23] | 1.3 [0.5 to 3.4] | 9.5 [3.8 to 23.8] | 1 [0.7 to 1.4]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 4 [0.7 to 23.8] | 4.9 [1.2 to 19.2] | 3.4 [0.8 to 13.3] | 3.3 [0.6 to 17] | 1.2 [0.5 to 2.7] | 14.7 [2.2 to 100.1] | 1.3 [0.6 to 2.8] | 3.7 [0.9 to 16.1] | 1.9 [0.8 to 4.4] | 8.8 [4.1 to 19.2] | 1 [0.7 to 1.4]

20. Secondary Outcome: Percentage of Participants With Seroresponse (4-Fold Rise) of Anti-norovirus GI.1 and GII.4 VLP IgA, IgG, and IgM Combined Using Pan-Ig ELISA
Description: as for outcome 15
Time Frame: I run: 7, 21, 28 days PD1, 7 and 28 days PD2; II run: 28, 152 and 365 days PD2 (up to Day 393)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
percentage of participants
  GI.1: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD1 | 88.9 [51.8 to 99.7] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GI.1: I Run:21 Days PD1 | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD1 | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 88.9 [51.8 to 99.7] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:7 Days PD2 | 100.0 [66.4 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [63.1 to 100.0] | 25.0 [3.2 to 65.1] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 100.0 [66.4 to 100.0] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: I Run:28 Days PD2 | 100.0 [66.4 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 25.0 [3.2 to 65.1] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 100.0 [66.4 to 100.0] | 11.1 [0.3 to 48.2] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:28 Days PD2 | 100.0 [66.4 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 14.3 [0.4 to 57.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 100.0 [66.4 to 100.0] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GI.1: II Run:152 Days PD2 | 87.5 [47.3 to 99.7] | 100.0 [59.0 to 100.0] | 100.0 [66.4 to 100.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 100.0 [66.4 to 100.0] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GI.1: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GI.1: II Run:365 Days PD2 | 66.7 [22.3 to 95.7] | 100.0 [59.0 to 100.0] | 100.0 [63.1 to 100.0] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 41.0] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 11.1 [0.3 to 48.2] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 7 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD1 | 66.7 [29.9 to 92.5] | 75.0 [34.9 to 96.8] | 80.0 [44.4 to 97.5] | 71.4 [29.0 to 96.3] | 0.0 [0.0 to 36.9] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 30.8] | 66.7 [29.9 to 92.5] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:21 Days PD1: number analyzed (Participants) | 9 | 8 | 10 | 8 | 8 | 8 | 10 | 8 | 8 | 8 | 7
  GII.4: I Run:21 Days PD1 | 55.6 [21.2 to 86.3] | 87.5 [47.3 to 99.7] | 80.0 [44.4 to 97.5] | 75.0 [34.9 to 96.8] | 0.0 [0.0 to 36.9] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 36.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD1 | 55.6 [21.2 to 86.3] | 87.5 [47.3 to 99.7] | 80.0 [44.4 to 97.5] | 75.0 [34.9 to 96.8] | 12.5 [0.3 to 52.7] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: I Run:7 Days PD2: number analyzed (Participants) | 9 | 7 | 10 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:7 Days PD2 | 66.7 [29.9 to 92.5] | 71.4 [29.0 to 96.3] | 80.0 [44.4 to 97.5] | 75.0 [34.9 to 96.8] | 12.5 [0.3 to 52.7] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GII.4: I Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 8 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: I Run:28 Days PD2 | 55.6 [21.2 to 86.3] | 85.7 [42.1 to 96.6] | 88.9 [51.8 to 99.7] | 75.0 [34.9 to 96.8] | 12.5 [0.3 to 52.7] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GII.4: II Run:28 Days PD2: number analyzed (Participants) | 9 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:28 Days PD2 | 66.7 [29.9 to 92.5] | 71.4 [29.0 to 96.3] | 88.9 [51.8 to 99.7] | 75.0 [34.9 to 96.8] | 14.3 [0.4 to 57.9] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 30.8] | 77.8 [40.0 to 97.2] | 0.0 [0.0 to 33.6] | 100.0 [63.1 to 100.0] | 0.0 [0.0 to 41.0]
  GII.4: II Run:152 Days PD2: number analyzed (Participants) | 8 | 7 | 9 | 8 | 7 | 8 | 10 | 9 | 9 | 8 | 7
  GII.4: II Run:152 Days PD2 | 50.0 [15.7 to 84.3] | 57.1 [18.4 to 90.1] | 66.7 [29.9 to 92.5] | 50.0 [15.7 to 84.3] | 14.3 [0.4 to 57.9] | 87.5 [47.3 to 99.7] | 10.0 [0.3 to 44.5] | 66.7 [29.9 to 92.5] | 11.1 [0.3 to 48.2] | 87.5 [47.3 to 99.7] | 0.0 [0.0 to 41.0]
  GII.4: II Run:365 Days PD2: number analyzed (Participants) | 6 | 7 | 8 | 7 | 7 | 8 | 10 | 9 | 9 | 7 | 7
  GII.4: II Run:365 Days PD2 | 33.3 [4.3 to 77.7] | 57.1 [18.4 to 90.1] | 62.5 [24.5 to 91.5] | 42.9 [9.9 to 81.6] | 14.3 [0.4 to 57.6] | 62.5 [24.5 to 91.5] | 10.0 [0.3 to 44.5] | 55.6 [21.2 to 86.3] | 22.2 [2.8 to 60.0] | 100.0 [59.0 to 100.0] | 0.0 [0.0 to 41.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and up to 365 Days after post dose 2 (Day 393)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg | Cohort A1-A4: Placebo | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort B: Placebo | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg | Cohort C: Placebo | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg | Cohort D: Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 1/10 | 0/9 | 0/9 | 0/9 | 1/10 | 2/10 | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/10 | 5/10 | 5/10 | 3/9 | 3/9 | 5/9 | 3/10 | 4/10 | 5/9 | 5/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg (N=10) | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg (N=10) | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=10) | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg (N=9) | Cohort A1-A4: Placebo (N=9) | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=9) | Cohort B: Placebo (N=10) | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=10) | Cohort C: Placebo (N=9) | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg (N=8) | Cohort D: Placebo (N=8)
Idiopathic central retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fractured right fibula (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bleeding following urologic surgery (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 5/5 mcg (N=10) | Cohort A2: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 15/15 mcg (N=10) | Cohort A3: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=10) | Cohort A4:Norovirus Bivalent GI.1/GII.4 VLP Vaccine 150/150mcg (N=9) | Cohort A1-A4: Placebo (N=9) | Cohort B: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=9) | Cohort B: Placebo (N=10) | Cohort C: Norovirus Bivalent GI.1/GII.4 VLP Vaccine 50/50 mcg (N=10) | Cohort C: Placebo (N=9) | Cohort D: Norovirus Bivalent VLP GI.1/GII.4 Vaccine 50/50 mcg (N=8) | Cohort D: Placebo (N=8)
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 3 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Capillary fragility (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mean cell haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Red cell distribution width increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.